CLINICAL TRIAL: NCT04420845
Title: Diabetes Self-Management Education with Sleep Hygiene
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was significantly delayed due to the COVID-19 pandemic. The PI has chosen not to conduct the study.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 239740
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2; Sleep Hygiene
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Hygiene | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Other)
  Interventions: Behavioral: Diabetes Self-Management and Support (DSMES) and Sleep Hygiene Education and Support (SHES)

INTERVENTIONS:
Behavioral: Diabetes Self-Management and Support (DSMES) and Sleep Hygiene Education and Support (SHES) — SHES outlines the importance of sleep for people with type 2 diabetes mellitus and provide practical information and guidance about sleep habits. Specifically, the focus will be on: avoiding consumption of caffeine, nicotine, alcohol; avoiding use of light emitting devices before bedtime; avoiding excessive intake of fluids or heavy meals before bedtime; promoting regulation of light, noise, and temperature in the bedroom; timing of and importance of exercise; maintaining consistent sleep and wake times; establishing a pre-bedtime routine; and managing stress.

SUMMARY:
This study will test whether adding sleep hygiene education and support to diabetes self-management education and support (DSMES) in diverse patients (African American, Hispanic, Pacific Islander, and Caucasian) with type 2 diabetes myelitis (T2DM) from rural UAMS Regional Programs clinics is more effective than DSMES alone. The specific aims for this study are:

* Aim 1A (Primary): Determine if this model improves blood glucose levels as measured by the HbA1c test in diverse adults with T2DM.
* Aim 1B: Determine the preliminary effectiveness of DSMES+SHES on sleep duration and sleep quality, blood pressure, fasting lipids, body mass index (BMI), self-management behavior, self-efficacy, diabetes-related distress, and diabetes-related quality of life in diverse adults with T2DM.
* Aim 2A: Determine the feasibility and acceptability of DSMES+ SHES when implemented with diverse adults with T2DM.
* Aim 2B: Determine the feasibility and acceptability of DSMES+ SHES implementation in Regional Programs clinics.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with type 2 diabetes
* Speak English

Exclusion Criteria:

* Received DSME in the past three years
* Have a condition that makes it unlikely they will be able to follow the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Change in mean HbA1c (NGSP%) from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  A Siemens analyzer will be utilized to calculate HbA1c (%) for each participant at each time point. Changes in the primary outcome measure will be assessed from baseline to post-intervention.

SECONDARY OUTCOMES:
Change in sleep duration from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  Self-reported sleep duration (hours slept) will be assessed using valid Behavioral Risk Factor Surveillance System survey items.
Change in sleep quality from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  The PROMIS® Short Form v1.0- Sleep Disturbance-4a scale will be used to assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep.This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep.
Change in mean blood pressure (systolic & diastolic, mmHg) from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  Blood pressure will be measured with a sphygmomanometer and stethoscope or digital blood pressure device with the participant seated and arm elevated.
Change in mean body mass index (BMI) from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  BMI will be collected by measuring participant height (without shoes) using a stadiometer, and by measuring participant weight (without shoes) using a calibrated digital scale. Participant weight and height will then be used to compute a continuous measure of BMI.
Change in mean total cholesterol (mg/dL) from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  Through finger prick blood collection, point of care tests will be used used to test total cholesterol using a commercial lipid panel kit and Cholestech LDX analyzer.
Change in mean low-density lipoproteins (LDL) (mg/dL) from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  Through finger prick blood collection, point of care tests will be used used to test LDL using a commercial lipid panel kit and Cholestech LDX analyzer.
Change in mean high-density lipoproteins (HDL) (mg/dL) from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  Through finger prick blood collection, point of care tests will be used used to test HDL using a commercial lipid panel kit and Cholestech LDX analyzer.
Change in mean triglycerides (mg/dL) from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  Through finger prick blood collection, point of care tests will be used used to test triglycerides using a commercial lipid panel kit and Cholestech LDX analyzer.
Change in diabetes self-management behaviors from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  The Summary of Diabetes Self-Care Activities (SDSCA) will be used to measure engagement in self-management activities. The SDSCA consists of 12 items to assess the self-reported frequency of performing diabetes self-care tasks, including testing blood sugar, following healthful eating plans, and exercising regularly.
Change in diabetes-related self-efficacy from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  The Diabetes Management Self-Efficacy Scale (DMSES) will be used to measure patient's confidence in managing their diabetes. The DMSES consists of 8 items to assess self-reported confidence in managing aspects of their diabetes. Items are scored on a 0-10 point scale, with higher scores indicating higher levels of self-efficacy.
Change in diabetes-related distress from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  The Problem Areas in Diabetes Scale (PAID)-5 will be used to measure diabetes distress. The PAID-5 consists of 5 items to assess self-reported diabetes-related emotional distress, including feeling scared or depressed. Items are scored on a 0-4 point scale, with higher scores indicating higher levels of distress.
Change in diabetes-related quality of life from baseline to 12 weeks post-intervention | Baseline and 12 weeks post-intervention
  The DAWN2 Impact of Diabetes Profile (DIDP) will be used to measure the perceived impact of diabetes on patients' quality of life. The DIDP consists of 6 items to assess self-reported impacts on quality of life, including physical health, financial situation, and relationships with others.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences Northwest, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No